CLINICAL TRIAL: NCT03366584
Title: The Effect of Co-administered β-Carotene, Vitamin D3, Zinc and Antenatal Steroid Therapy on Hyaline Membrane Disease and Feeding Intolerance in Premature Neonates
Brief Title: The Effect of β-Carotene, Vitamin D3 and Zinc on Hyaline Membrane Disease and Feeding Intolerance in Premature Neonates
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Yuyun Lisnawati, dr, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 190/2016
Record Dates: First submitted 2017-12-03; First posted 2017-12-08 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Hyaline Membrane Disease; Necrotizing Enterocolitis of Newborn
MeSH Terms: conditions — Hyaline Membrane Disease | interventions — beta Carotene; Cholecalciferol; Zinc; picolinic acid; Dexamethasone

STUDY DESIGN:
Intervention Model Description: The research will be held in Cipto Mangunkusumo General Hospital. Each participant of each group will be given dexamethasone 2x6 mg intravenous for 2 days which aims to support lung maturation followed by planned delivery within 1 week due to indication of maternal or fetal. The maternal dan cord blood sample are obtained for zinc, vitamin A and 25(OH)D levels examinations. Randomly, subjects will be divided into 2 groups which are group who is given the oral beta-carotene 25,000 IU, oral vitamin D3 50,000 IU and oral zinc 50 mg/day for 3 days, and group who is not given the intervention. After the premature neonates was born, observation will be done for maximum period of 4 weeks. The presence and severity of HMD and feeding intolerance or NEC will be recorded.
Who Masked: Outcomes Assessor
Masking Description: The neonates outcomes, hyaline membrane disease and feeding intolerance, will be assessed for maximum period of 4 weeks by doctor who in charge in NICU. They are outside the research team and blind to maternal treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): * beta carotene 25,000 IU
  * vitamin D3 50,000 IU
  * zinc 50 mg
  * dexamethasone 6 mg
  Interventions: Dietary Supplement: Beta carotene; Dietary Supplement: Vitamin D3; Dietary Supplement: Zinc; Drug: Dexamethasone
- Control (Active Comparator): dexamethasone 6 mg
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Dietary Supplement: Beta carotene — Beta carotene 25,000 IU
  Arms: Intervention
Dietary Supplement: Vitamin D3 — Vitamin D3 50,000 IU
  Other Names: Cholecalciferol
  Arms: Intervention
Dietary Supplement: Zinc — Zinc 50 mg
  Other Names: Zinc picolinate
  Arms: Intervention
Drug: Dexamethasone — Dexamethasone 6 mg

SUMMARY:
Hyaline membrane disease, now commonly called respiratory distress syndrome (RDS), and feeding intolerance, which can lead to necrotizing enterocolitis (NEC), are two key morbidities found in premature neonates which resulted in high mortality rate in Indonesia. Cochrane meta-analysis proved that antenatal steroid therapy can reduce the morbidity and mortality rate of premature neonates. But there is still different outcomes and severity of disease in preterm newborn receiving the same dose of antenatal steroid therapy. This raises questions whether there are other factors influencing the development and maturity of lung and gut in preterm newborn, aside from steroid therapy. Vitamin A, D and zinc are already known for their function in fetal lung and gut development. To our best of knowledge, no study has evaluated the effect of these vitamins levels on HMD and feeding intolerance in premature neonates. Therefore, the aim of this study want to evaluate the effect of antenatal steroid therapy versus co-administered β-carotene, vitamin D3, zinc and antenatal steroid therapy on the presence and severity of HMD and feeding intolerance in premature neonates.

DETAILED DESCRIPTION:
This study is a randomized controlled trial and held in Cipto Mangunkusumo Hospital.

Pregnant women 28-34 weeks of gestational age, who fulfill the inclusion criteria, divide into two groups. Subjects from both groups receive the hospital protocol of preterm birth, 4 doses of 6 mg of dexamethasone, intravenous 12 hours apart to support lung maturation. Subjects in intervention group receive oral single-dose beta-carotene 25,000 IU, oral single-dose vitamin D3 50,000 IU and oral zinc 50 mg/day for 3 days. The maternal dan cord blood sample are obtained for zinc, vitamin A and 25(OH)D levels before and after intervention. After the premature neonates was born, observation will be done for maximum period of 4 weeks. The presence and severity of HMD and feeding intolerance or NEC will be recorded. Neonates showing any signs of HMD and/or abdominal distension will need to undergo additional chest/abdominal x-ray procedures.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who has preterm birth in 28-34 weeks gestational age

Exclusion Criteria:

* Multiple pregnancy
* Drug allergy
* Fetal congenital malformation
* Maternal gestational diabetes mellitus

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Hyaline membrane disease | 1,5 years
  The presence and severity of RDS (HMD) will be noted, according to chest X-ray result

SECONDARY OUTCOMES:
Feeding Intolerance | 1,5 years
  The presence and severity of necrotican enterocolitis will be noted, according to abdominal x-ray result

CONTACTS AND LOCATIONS:
Overall Officials: Yuyun Lisnawati, Study Chair — Persahabatan General Hospital
Locations (1):
- Cipto Mangunkusumo General Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
The research findings will be disseminated via publication of results